CLINICAL TRIAL: NCT00666575
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Actual Use Study of the Safety and Tolerability of Gabapentin 500 mg in a Potential OTC Population
Brief Title: A Study of the Safety of Gabapentin in a Potential Over-the-Counter Population With Occasional Sleeplessness
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A9451146
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2008-04

CONDITIONS: Transient Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gabapentin (Experimental)
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — Gabapentin 500 mg oral capsule 30 minutes prior to bedtime for 28 days
  Arms: Gabapentin
Drug: Placebo — Matched placebo oral capsule 30 minutes prior to bedtime for 28 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety of gabapentin, as compared to placebo, in a potential over-the-counter population with reports of occasional sleeplessness

ELIGIBILITY:
Inclusion Criteria:

* Subjects >/= 12 years of age who reported occasional sleeplessness in month prior to screening

Exclusion Criteria:

* Females who were pregnant or breastfeeding

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2105 (Estimated)
Dates: Start 2004-12; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Day 45

SECONDARY OUTCOMES:
Pulse and Blood Pressure | Day 45
Subjective proportion of nights having difficulty sleeping | Day 45
Subjective Sleep Latency | Day 45
Subjective Wake After Sleep Onset | Day 45
Subjective Number of Awakenings | Day 45
Subjective Total Sleep Time | Day 45
Subjective Assessment of Sleep Quality | Day 45
Subjective Assessment of Ease of Awakening | Day 45
Subject Global Evaluation | Day 45
Pittsburg Sleep Quality Index | Day 45

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (20):
- United States (20):
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Beverly Hills, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, DeLand, Florida
  - Pfizer Investigational Site, New Port Richey, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Boise, Idaho
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Santa Fe, New Mexico
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, West Jordan, Utah

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9451146&StudyName=A%20Study%20of%20the%20Safety%20of%20Gabapentin%20in%20a%20Potential%20Over-the-Counter%20Population%20with%20Occasional%20Sleeplessness